CLINICAL TRIAL: NCT02281721
Title: Prospective, Observational, Multi-Center, Single-Arm, Consecutive Enrollment, Post-Marketing, International Registry of the Surpass™ Flow Diverter in Intracranial Arteries
Brief Title: Surpass Flow Diverter for Intracranial Aneurysms: SURMOUNT Registry Data Collection
Status: Terminated | Type: Observational
Why Stopped: Internal decision
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: T4029
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single Group; Surpass Flow Diverter(s): Individuals using the Surpass Flow Diverter(s)
  Interventions: Device: Surpass Flow Diverter(s)

INTERVENTIONS:
Device: Surpass Flow Diverter(s) — Endovascular placement of a Surpass Flow Diverter(s) for the treatment of an intracranial aneurysm(s)

SUMMARY:
The purpose of this observational post-marketing registry will be to collect and analyze safety, effectiveness, and quality of life outcomes, during and after treatment with the Surpass Flow Diverter. Health Economics assessments (cost data) will also be collected and analyzed.

DETAILED DESCRIPTION:
This will be a prospective, observational, multi-center, single-arm, post-marketing, international registry with consecutive enrollment of a minimum of 150 patients treated with the Surpass Flow Diverter in accordance with the standard of care at up to 30 registry sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to be treated with a Surpass Flow Diverter(s) will be eligible to participate in this registry. Patients will be enrolled on a consecutive basis.

Exclusion Criteria:

* This is a standard of care registry. Patients should be excluded if standard of care at a given site is such that they are not eligible for treatment with a Surpass Flow Diverter(s).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For the primary endpoint, the evaluable patient population will consist of all individuals treated with the Surpass Flow Diverter(s) who have provided consent, and who have completed their 12 month follow-up assessment.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-03-18 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Primary effectiveness based on the proportion of patients with 100% aneurysm occlusion | 12 months
  The proportion of patients with 100% aneurysm occlusion, based on an assessment of each patient's imaging at 12 months (± 180 days) post-procedure, and stratified across four aneurysm categories.

SECONDARY OUTCOMES:
Technical success assessed by deployment of the device with complete coverage of the aneurysm neck | Peri-procedural
  Successful deployment of the device with complete coverage of the aneurysm neck.

OTHER OUTCOMES:
Safety outcomes assessed by neurological adverse events | Up to 5 years
  Neurological adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A Brouwer, MD, Principal Investigator — Karolinska Hospital
Locations (19):
- AZ groeninge, Kortrijk, Belgium
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turun yliopistollinen keskussairaala, Turku
- France (4):
  - Hopital Jean Minjoz, Besançon
  - APHP - Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Fondation Rothschild, Paris
  - Hopital Bretonneau, Tours
- Germany (3):
  - Freiburg University Hospital, Freiburg im Breisgau
  - Klinikum Kassel, Kassel
  - Universitätsmedizin Mannheim, Mannheim
- Italy (2):
  - San Martino Hospital, Genova
  - Neuroradiologia Azienda ILSS9, Treviso
- Radboudumc, Nijmegen, Netherlands
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander
- Karolinska University Hospital in Solna, Department of Neuroradiology, Stockholm, Sweden
- United Kingdom (3):
  - Queen's Hospital of Romford, NHS Barking, Havering and Redbridge University Hospitals Trust, Romford, Essex
  - Queen Elizabeth Hospital, Birmingham
  - The Walton center, Liverpool